CLINICAL TRIAL: NCT04775095
Title: BRAF V600-mutated Lung Carcinoma Treated With the Combination of Dabrafenib-trametinib: a Retrospective Evaluation (Secondary Data Use Study of Dabrafenib-Trametinib in "Real Life" for Non-Small Cell Lung Cancer With a BRAF V600 Mutation)
Brief Title: BRAF V600-mutated Lung Carcinoma Treated With the Combination of Dabrafenib-trametinib: a Retrospective Evaluation
Acronym: BLaDE
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: IFCT-2004
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Non Small Cell Lung Cancer; BRAF V600 Mutation
Keywords: Non-Small Cell Lung Cancer; BRAF V600 Mutation; Real-world study; IFCT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BLaDE cohort will evaluate overall survival (OS), real world progression-free survival (PFS), best response and duration of treatment in patients with advanced, metastatic Non-Small Cell Lung Cancer (NSCLC) harboring BRAF V600E or non E mutation who received dabrafeninb-trametinib combination or not. Subsequent or previous treatments (treatments delivered after or before dabrafeninb-trametinib combination will be recorded). Those outcomes will be correlated to clinical, pathological, and radiological characteristics of patients.

DETAILED DESCRIPTION:
The braf gene (V Raf murine sarcoma viral oncogene homolog, long arm of chromosome 7q3) codes for a protein (serine / threonine kinase) which regulates the signaling pathway RAS - RAF - MEK - ERK playing an important role in the proliferation processes, cell survival, angiogenesis, cell invasion and migration.

When activated by mutations, BRAF phosphorylates MEK to promote cell growth, proliferation and survival. In non-small cell lung cancer (NSCLC), BRAF mutations are found in 1-2% of cases. BRAF mutations are distinguished by kinase activity and their signaling via the mitogen-activated kinase (MAPK) pathway. BRAF V600 mutations, class I, signal as monomers with or without activated RAS. BRAF non-V600 are classified as either class II that signal as dimmers when RAS as activated or class III with impaired kinase activity but increased MAPK pathway signaling. The most frequent mutation in NSCLC (50% of cases) is the V600E mutation (glutamate / valine substitution, codon 600 of exon 15) which is activating (others mutations: G469A and D594G, respectively 39% and 11% of cases). One phase II trial demonstrated that the dabrafenib-trametinib combination had significant anti-tumor activity in terms of response rate, PFS in patients with a NSCLC with the BRAF V600E mutation, pretreated or not. In this multicentre non-randomized phase II open label study, a dabrafenib-trametinib combination was tested in 59 previously treated patients with metastatic stage IV BRAF V600E mutated NSCLC with documented progression after at least one prior platinum based chemotherapy. Overall response rate (ORR) was 63.2% (95% CI: 49.3 to 75.6%), median PFS was 9.7 months (95%CI 6.9-19.6). In the cohort of patients previously untreated (n=36) and treated with first line dabrafenib-trametinib combination, the investigator-assessed confirmed ORR was 64% (95% CI 46-79 %), the median investigator assessed PFS was 10.9 months (95CI:7-16.6) and the 6 month-PFS was 72% (53-84%) respectively.

At the last ASCO conference 2020, the data have been updated. In cohorts of untreated and previously treated patients, the ORR was 63.9% (95CI 46.2-79.2) and 68.4% (95CI 54.8, 80.1), median PFS 10.8 months (95CI 7.0-14.5) and 10.2 months (95CI: 6.9-16.7). Median OS was 17.3 months (95% CI: 12.3-40.2; 3 years OS: 40%) and 18.2 months (95% CI: 14.3-28.6; 3 years OS: 33%) with 14/36 and 11/57 patients alive in treatment naïve and pretreated patients respectively.

The dabrafenib-trametinib combination had European authorization since 2017. In January 2020, the French Transparency Committee validated its possible use in second line in current practice, after failure of a first therapeutic line (whatever its nature) but only for BRAF V600E mutations. Clinical outcomes data on BRAF-mutated V600 NSCLC patients treated in routine practice by dabrafenib-trametinib combination is limited with only retrospective studies including few patients.

The primary objective of this retrospective multicenter observational study is to describe, in real world, the characteristics and evolution of NSCLC patients with a BRAF V600 E mutation treated with the dabrafenib-trametinib combination regardless of the line of treatment. Also, this retrospective multicenter observational will describe in real world, the characteristics, treatment and evolution of NSCLC patients with a BRAF V600 non E mutation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed extensive stage NSCLC
* Presence of BRAF V 600 E or non E mutation diagnosed on tumor sample and/or on liquid biopsy (co mutations allowed) between 01/01/2016 and 31/12/2019
* Patients who received at least one dose of treatment with dabrafenib-trametinib combination (whatever the treatment line)
* NSCLC BRAF V600 patients who have not received the dabrafenib-trametinib combination will be included for the collection of clinical and demographic data, treatments received and OS
* Patients who were informed about the study and do not refused for their data to be collected and used
* Age > 18 years

Exclusion Criteria:

* Patients harboring a non V600 BRAF mutation
* Patients enrolled in a clinical trial assessing treatment with dabrafenib-trametinib combination
* Explicit refusal by the patient to collect his or her data
* Patients under curatorship or guardianship
* Unable to obtain data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with histologically or cytologically confirmed extensive stage NSCLC with BRAF V600 (E or non E) mutation diagnosed on tumor sample and/or on liquid biopsy (co mutations allowed) between 01/01/2016 and 31/12/2019
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) at 12 months in non-small cell lung cancer (NSCLC) BRAF V600E-mutated patients receiving the combination of dabrafenib-trametinib as second line or more treatment | 12 months
  OS will be determined as the time from the first dose of treatment with dabrafenib-trametinib to death from any cause

SECONDARY OUTCOMES:
OS at 18 and 24 months and median OS in NSCLC BRAF V600E-mutated patients receiving the combination of dabrafenib-trametinib as second line or more treatment | 18 and 24 months
  OS will be determined as the time from the first dose of treatment with dabrafenib-trametinib to death from any cause
OS at 12, 18 and 24 months and median OS in NSCLC BRAF V600E-mutated patients receiving the combination of dabrafenib-trametinib as first-line treatment | at 12, 18 and 24 months
  OS will be determined as the time from the first dose of treatment with dabrafenib-trametinib to death from any cause
OS at 12, 18 and 24 months and median OS in NSCLC BRAF V600E-mutated patients regardless of the treatment received | at 12, 18 and 24
  OS will be determined as the time from the first dose of treatment with dabrafenib-trametinib to death from any cause
OS at 12, 18 and 24 months and median OS in NSCLC BRAF V600E-mutated patients not treated by the combination of dabrafenib-trametinib, according to the treatment and the line received | at 12, 18 and 24
  OS will be determined as the time from the first dose of treatment with dabrafenib-trametinib to death from any cause
OS at 12 months and median OS in NSCLC BRAF V600 non E-mutated patients according to the treatment and the line received | at 12 months
  OS will be determined as the time from the first dose of treatment with dabrafenib-trametinib to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard AULIAC, Dr, Study Chair — Créteil -CHI; Aurélie SWALDUZ, Dr, Study Chair — Lyon - CLCC
Locations (2):
- France (2):
  - Créteil - CHI, Créteil
  - Lyon - CRLCC, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: IFCT website — https://www.ifct.fr/etudes-cliniques/141-ifct-2004